CLINICAL TRIAL: NCT04214912
Title: Yeur-Hur Lai, PhD, RN, School of Nursing, College of Medicine, National Taiwan University
Brief Title: Personalized Survivor Care Plan for Oral Cancer Patients-Effects on Physical-Psychological Functions and Return-to-Work
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201703103RINC
Record Dates: First submitted 2018-11-27; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Oral Cancer
Keywords: Oral Cancer; Intervention; Return to work
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Intervention Model Description: There are various models of SCP, in general, the primary care physician model or nurse-led model are generally being recognized for effective detecting patients' distress and recurrences, effective coordination and communication, and taking SCP as standard cancer care. In Taiwan, we take a large number of advanced OC patients, it is important to integrate the SCP but also need to concern about the limited time in busy OPD clinics and patients' differences because of various physical or psychological conditions and needs. PSCP-OC will include two major modules: General & Personalized Modules.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was not fully blinded; however, the group allocation was concealed from the patient and primary researcher until after baseline assessments were completed. A primary researcher obtained patient consent, collected self-reported assessments, and if the patients were randomized to intervention group, the intervention trainer explained the exercise program to participants. The study statistician and data managers remained blinded at all times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General module (No Intervention): General module will serve as a "roadmap plan" which will cover the most common problems and major issues related to current and future treatments, side effects, psychological distress, daily function and physical condition. The contents will be developed based on empirical review, our current research findings in Taiwan, OC health care experts' suggestions.
- Personalized module (Experimental): Personalized Survivor Care Plan (PSCP) will deliver based on what we assess or interview about patients' distress, concerns and care needs in each interview or/and assessment. We will assess OC patients of the above items by valid assessment tools. For the factors or concerns about RTW assessment, we will develop and test a modified instrument for the study purpose. For each assessment, the computer -assisted assessment will help the OC educator to immediately catch the patients care distress and care needs. It will provide the direction for caring of their personalized distress, concerns and needs.
  Interventions: Combination Product: Personalized Survivor Care Plan (PSCP)

INTERVENTIONS:
Combination Product: Personalized Survivor Care Plan (PSCP) — Based the above literature review and our previous 10 years' efforts in OC patients' distress and care needs survey, we categorize OC patients' distress and needs into 6 major dimensions (1) symptoms management and dysfunction prevention (different kind of symptom, such as swallowing difficulty, eating difficulty, speaking difficulty, difficulty in opening mouth/trismus, shoulder dysfunction, mucositis, pain, fatigue, etc), (2) enhancing physical function (exercise skills, types for major parts of muscle training), (3) Confronting and dealing with psychological distress (fear, anxiety, depression, uncertainty), (4) nutrition assessment and counseling, (5) Social connection and RTW counseling (attitudes and skills for returning to work), and (6) overall needs assessment and supports.
  Arms: Personalized module

SUMMARY:
Background: Due to the complex treatment modalities and long-term side effects, oral cancer (OC) patients might suffer from psychological and physical distress and be unable to return to work (RTW).

Purposes: This is a two-phase study. First, the investigator aims to validate a scale about OC patients' perception of RTW and identify those concerns in RTW. Second, the investigator aims to (1) develop the contents of a "Personalized Survivorship Care Plan- Oral Cavity Cancer (PSCP-OC)" and (2) examine the short and long-term effects of PSCP-OC on patients' physical function (symptoms, muscle strengths, fitness, nutrition status), psychological distress (depression, fear of cancer recurrence) and RTW.

Method: First phase, the investigator will modify and validate the "Illness Perception Questionnaire (IPQ)" with adding the head and neck cancer specific items (modified IPQ-mHN) to assess the barriers of RTW in OC patients. The investigator will recruit 300 subjects in this phase to test the IPQ-mHN psychometrics. The second and third year will develop and test the PSCP-OC intervention. Eligible subjects will be (1) newly diagnosed OC patients with surgery, and (2) who are at work in time of diagnosis. A stratified randomization by cancer stage would be conducted. Both groups will receive baseline assessment before first intervention. PSCP-OC is a 6-month intervention which includes two parts: General module and Personalized module (150 subjects for each group). Ex group will receive the first PSCP-OC before discharge and 3 times face-to-face PSCP-OP once a month in the first three month after discharge and 3 times telephone physical-psycho-education interventions in month 4-6. Control group will receive regular and cancer case manager cares for 6 months. Each group will be followed for 12 months and assess of their outcomes at 6 time points: baseline (pre-discharge) and 1, 3, 6, and 12 months after surgery. Outcomes will be evaluated by physical distress, muscle strength, nutrition status, and length of time of RTW since completion of last major treatment. Results would be analyzed mainly by GEE. IRB approval will be received before the RCT.

Expected Outcome: Expecting to develop a scale to identify those barriers preventing OC patients' RTW and further to test the PSCP. A promising result will further apply into clinical care to prevent or decrease the potential declined physical and psychological functions, increase their strength and help them RTW.

DETAILED DESCRIPTION:
Supportive Care has been proved to not only increase patients' life quality but also their survival time. An influential randomized control study published on the New England Journal of Medicine (Temel et al., 2010) found that the early palliative (supportive) care could significantly improve patients' QOL and median survival time (11.6 month vs. 8.9 months) in a 151 metastatic NSCLC patients. This study strongly supports our clinical care needs and scientific assumption that effective and continuous supportive care is needed in advanced OC patients.

However, in Taiwan, there is no insurance paying for supportive care in both inpatient and particularly in OPD (only pay for treatment and physician fee). In order to meet patients' care need and concerning the reality of our medical payment system, the investigator aims to develop a systematic well-planed and efficient survivor care plan (SCP), with taking consideration of OC patients/survivors' personal care needs across different cancer process.

Survivorship Care Plan (SCP) Cancer survivor is defined as "any patient who has been diagnosed with cancer and continues through their lifespan(NIH, 2014)". One of the most important reports about survivorship care and content of care has been reported by Institute of Medicine (IOM, 2006). According to IOM, the essential component of survivorship care includes "communication and coordination of care, prevention and detection of recurrence, assessment and management of treatment/disease related distress or late effects. A well-designed survivor care plan (SCP) has been viewed as an important communication tool to improve transitions of care for cancer patients. Increasing attentions and reports have been found about the values of SCP from Office of Cancer Survivorship, and American Society of Clinical oncology (Mayer, 2014) and strongly suggest to use SCP in clinical cancer practice to increase the care quality and long-term cancer survivors' quality of life.

There are various models of SCP, in general, the primary care physician model or nurse-led model are generally being recognized for effective detecting patients' distress and recurrences, effective coordination and communication, and taking SCP as standard cancer care. In Taiwan, the investigator takes a large number of advanced OC patients, it is important to integrate the SCP but also need to concern about the limited time in busy OPD clinics and patients' differences because of various physical or psychological conditions and needs.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed operable oral cavity cancer patients with at least neck dissection
* patients has work at time of diagnosis

Exclusion Criteria:

* primary unknown
* conscious unclear
* recurrence or with bone meta

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in University of Washington - Quality of Life (UW-QoL) | We will assess patients' the changes of outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital)
  It is characterized of its simplicity and developed to quickly assess head and neck cancer patients' health related QOL. Four versions have been developed since 1993 (Hassan & Wymuller, 1993; Weymuller, Alsarraf, Yueh, Deleyiannis, & Coltrera, 2001). The current version, UW-QOL version 4 contains 12 items that to assess 12 domains of QOL in head and neck cancer patients, and each domain is scored from 0-100 with the higher scores indicating better function (Roger et al., 2002). It has been translated into Chinese and tested for its psychometrics in our previous head and neck cancer populations in Taiwan (Lee et. al., 2018).
Changes in Hospital Anxiety & Depression Scale (HADS) | We will assess patients' the changes of outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital)
  The severity of cancer patients' anxiety and depression will be measured by the self-reported HADS. The 14 items of HADS consists of two subscales, include 7 items anxiety and 7 items depression. The score of all items ranges from 0 (not at all) to 3 (always) and the total score of each subscale are ranged from 0 to 21 with a higher score indicating a higher level of anxiety or depression. Satisfactory psychometrics of the HADS has been shown in cancer populations in Taiwan (Chen et al., 2000).
Changes in Illness Perception Questionnaire (IPQ) - the head and neck cancer specific items (modified IPQ-mHN) | We will assess patients' the changes of outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital)
  The questionnaire was originally developed from Broadbent, Petrie, Main and Weinman (2006) to measure patients' perception about their illness and it has proved to have good psychometric characteristics. The IPQ was further modified by Grunfeld. Low, and Cooper (2010) to assess cancer patients' perception about the impacts of cancer and its treatments on their work. Concerning about part of the purposes of this study is to examine OC patients' concerns, perception and barriers of their RTW and further use it to a wider range of HNC patients, we will therefore add head and neck cancer specific items to become IPQ-mHN to fit into different types of HNC and also OC patients. The 26 item IPQ-M was a 7-point Likert's scale with 0 to 7 scoring and the higher the sum scores (0-119) indicates more concerns or barriers about RTW.
Changes in Fear of Recurrence Questionnaire (FoR) | We will assess patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital)
  The FoR-C is a Chinese version of the original FoR questionnaire. The FoR questionnaire consists of six statements with a five-point response scale from not at all (1), a little, sometimes (2), a lot , and all the time) and one statement with a response scale from 0 (not at all) to 10 (a great deal). The summary of FoR ranges from 6 to 40. Higher score indicates a higher level of fear of recurrence. The significance of the FoR was indicated by patients' responses 'a lot' or 'all the time' for the first six statements and the score of 7-10 for the last item, in which case. Current study will use the same approach to determine the cut-off point of the FoR.
Changes in Exercise and Muscle Power | We will assess patients' the changes of outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital)
  This measures has been applied in PI's currently head and neck study and early stage lung cancer follow up study. Muscle strength and endurance we will use grip strength meter to measure the strength of right and left upper limbs; and will use microFET 2 to measure the strength of right and left hip flexor muscle. Both grip strength meter and microFET 2 provided good reliability and validity for measuring muscle strength in the past studies (Schaubert & Bohannon, 2005). First, patients will be asked to stand up, put arms by sides, and hold the meter to make a fist with maximal force for two times to record upper limbs strength. Secondly, patients will be seated on the chair. The researcher will put the microFET 2 on the upper edge of knee, and then let patient maintain the thigh raise for four seconds to record the strength of right and left hip flexor muscle.
Changes in Brief Supportive Care Needs Survey (SCNS-ST9) | We will assess patients' the changes of outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T6 = 1, 3, 6, and 12 months after discharge from hospital)
  The unmet needs of lung cancer patient will be measured by 9 items SCNS. It consists of 5 domains, include psychological, health system and information, daily living, patient care and sexuality domain. Response options "No need, not applicable (1); No need, satisfied (2); Low need (3); Moderate need (4); High need (5). The sum of item scores within each domain will be calculated and transformed to a standardized score from 0 to 100, with higher scores indicating more unmet needs (Girgis et al, 2011). The Chinese SCNS34 has acceptable psychometric properties in previous lung cancer studies (Liao et al., 2011; Shun et al., 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Yeur-Hur Lai, Professor, Study Chair — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- Otorhinolaryngology Department, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Hassan SJ, Weymuller EA Jr. Assessment of quality of life in head and neck cancer patients. Head Neck. 1993 Nov-Dec;15(6):485-96. doi: 10.1002/hed.2880150603. PMID 8253555
- [Background] Weymuller EA Jr, Alsarraf R, Yueh B, Deleyiannis FW, Coltrera MD. Analysis of the performance characteristics of the University of Washington Quality of Life instrument and its modification (UW-QOL-R). Arch Otolaryngol Head Neck Surg. 2001 May;127(5):489-93. doi: 10.1001/archotol.127.5.489. PMID 11346422
- [Background] Rogers SN, Lowe D, Fisher SE, Brown JS, Vaughan ED. Health-related quality of life and clinical function after primary surgery for oral cancer. Br J Oral Maxillofac Surg. 2002 Feb;40(1):11-8. doi: 10.1054/bjom.2001.0706. PMID 11883963
- [Background] Lee YH, Lai YH, Yueh B, Chu PY, Chen YJ, Chen SC, Wang CP. Validation of the University of Washington Quality of Life Chinese Version (UWQOL-C) for head and neck cancer patients in Taiwan. J Formos Med Assoc. 2017 Apr;116(4):249-256. doi: 10.1016/j.jfma.2017.01.002. Epub 2017 Feb 15. PMID 28214178
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Chen ML, Chang HK, Yeh CH. Anxiety and depression in Taiwanese cancer patients with and without pain. J Adv Nurs. 2000 Oct;32(4):944-51. PMID 11095234
- [Background] Grunfeld EA, Low E, Cooper AF. Cancer survivors' and employers' perceptions of working following cancer treatment. Occup Med (Lond). 2010 Dec;60(8):611-7. doi: 10.1093/occmed/kqq143. Epub 2010 Sep 20. PMID 20855546
- [Background] Schaubert KL, Bohannon RW. Reliability and validity of three strength measures obtained from community-dwelling elderly persons. J Strength Cond Res. 2005 Aug;19(3):717-20. doi: 10.1519/R-15954.1. PMID 16095431
- [Background] Girgis A, Lambert S, Lecathelinais C. The supportive care needs survey for partners and caregivers of cancer survivors: development and psychometric evaluation. Psychooncology. 2011 Apr;20(4):387-93. doi: 10.1002/pon.1740. Epub 2010 Apr 5. PMID 20878835
- [Background] McElduff, P., Boyes, A., Zucca, A., & Girgis, A. (2004). Supportive Care Needs Survey: A guide to administration, scoring and analysis. Newcastle: Centre for Health Research & Psycho-oncology.
- [Background] Liao YC, Liao WY, Shun SC, Yu CJ, Yang PC, Lai YH. Symptoms, psychological distress, and supportive care needs in lung cancer patients. Support Care Cancer. 2011 Nov;19(11):1743-51. doi: 10.1007/s00520-010-1014-7. Epub 2010 Oct 15. PMID 20949362
- [Background] Shun SC, Yeh KH, Liang JT, Huang J, Chen SC, Lin BR, Lee PH, Lai YH. Unmet supportive care needs of patients with colorectal cancer: significant differences by type D personality. Oncol Nurs Forum. 2014 Jan 1;41(1):E3-11. doi: 10.1188/14.ONF.E3-E11. PMID 24368251
- [Result] National Institutes of Health (NIH). About cancer survivorship. Available at: http://cancercontrol.cancer.gov/ocs/about/mission.html. Accessed May 30, 2014.
- [Result] Institute of Medicion (IOM). from cancer patient to cancer survivor-lost in transition. Washington, DC: The National Academies Press; 2006. Report no:0-309-09595-6. Available at: http:// www.iom.edu/reports/2005/from-cancer-patient-to-cancer-survivor-lost-in-transition.aspx.
- [Result] American College of Surgeons Commission on Cancer Cancer Program Standards, Version 1.2.1:ensuring Patient-Centered Care. Available at: http://deainfo.nci.nih.gov/advisory/pcp/archive/pcp00-01rpt/PCPvideo/voices_files/pcpanel.html. Accessed December 29, 2014.
- [Result] Mayer DK, Nekhlyudov L, Snyder CF, Merrill JK, Wollins DS, Shulman LN. American Society of Clinical Oncology clinical expert statement on cancer survivorship care planning. J Oncol Pract. 2014 Nov;10(6):345-51. doi: 10.1200/JOP.2014.001321. Epub 2014 Oct 14. PMID 25316025